CLINICAL TRIAL: NCT01601210
Title: Placebo-Controlled Dose-Ranging Trial of Creatine Augmentation for Adolescent Females With Treatment-Resistant Major Depressive Disorder: a Magnetic Resonance Spectroscopy Study
Brief Title: Dose-Ranging Trial of Creatine Augmentation for Adolescent Females With Treatment-Resistant Major Depressive Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Perry Renshaw (Other)
Responsible Party: Sponsor-Investigator, Perry Renshaw, MD, PhD, MBA, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00055231
Record Dates: First submitted 2012-04-17; First posted 2012-05-17 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Creatine monohydrate or placebo
- 2 grams of creatine (Active Comparator)
  Interventions: Drug: Creatine monohydrate or placebo
- 4 grams of creatine (Active Comparator)
  Interventions: Drug: Creatine monohydrate or placebo
- 10 grams of creatine (Active Comparator)
  Interventions: Drug: Creatine monohydrate or placebo

INTERVENTIONS:
Drug: Creatine monohydrate or placebo — Placebo, 2g, 4g, and 10g of creatine monohydrate

SUMMARY:
The purpose of this study is to see if creatine, which is a naturally occurring chemical in the body, is effective for treating Major Depressive Disorder (MDD) in female teenagers.

The primary hypothesis is that compared to placebo, 2g, 4g, and 10g of creatine monohydrate for eight weeks will be associated with a significant increase in brain phosphocreatine (PCr) concentrations.

DETAILED DESCRIPTION:
The purpose of this study is to see if creatine, which is a naturally occurring chemical in the body, is effective for treating Major Depressive Disorder (MDD) in female teenagers. Creatine may have effects of interest in the brain. The reason for the MRI component of this study is to learn about new ways to see inside the brain. The investigators will use magnetic fields and radio waves to look at the brain and chemicals in the brain. The investigators hope that this technique will have medial use in the future.

The primary hypothesis is that compared to placebo, 2g, 4g, and 10g of creatine monohydrate for eight weeks will be associated with a significant increase in brain phosphocreatine (PCr) concentrations. A secondary hypothesis is that decreased depressive symptoms measured with the Children Depression Rating Scale-Revised (CDRS-R) and Montgomery Asberg Depression Rating Scale (MADRS) will be reciprocally correlated with increased β-NTP concentrations.

ELIGIBILITY:
Inclusion criteria:

* Participants must be female.
* Participants must be able to grant informed consent (age > 18), or parent/guardian permission plus participant assent (age < 18).
* Participants must meet DSM-IV criteria for MDD, with current mood state depressed for > 2 weeks.
* Participants must be between the ages of 13 and 21.
* Current CDRS-R raw score of > 40 or MADRS score > 25; and CGI-S score > 4.
* Participants may be enrolled in individual and/or group psychotherapy, if it has been ongoing for at least 8 weeks.
* Participants must have been in treatment with an SSRI for at least 8 weeks, the last 4 of which were at a dosage of > or equal to 20 mg per day of fluoxetine or its equivalent, e.g. 20 mg per day of paroxetine, 20 mg citalopram, 10 mg escitalopram, or 100 mg sertraline. If the participant attempted, but could not tolerate, a dose comparable to 20 mg fluoxetine, they will be considered eligible.

Exclusion criteria:

* Unstable co-morbid medical, neurological, or psychiatric disorder.
* Current DSM-IV criteria for substance abuse or dependence (excepting nicotine/cigarettes).
* Clinically significant suicidal or homicidal risk.
* Pre-existing renal disease.
* Proteinuria on baseline urinalysis testing.
* Treatment with antiepileptic drugs, antipsychotic drugs, or lithium.
* Pregnancy or breastfeeding.
* Sexually active and unwilling to practice contraception during the study.
* Contraindication to magnetic resonance imaging (e.g. ferromagnetic implant or claustrophobia)
* History of hypersensitivity to creatine.
* History of a previous failed therapeutic trial of creatine.
* Participants may be outpatients or inpatients, but incarcerated persons will be excluded because this study is not approved for "Research Involving Prisoners."

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Brain PCr concentrations | 8 weeks
  The primary hypothesis is that compared to placebo, 2g, 4g, and 10g of creatine monohydrate for eight weeks will be associated with a significant increase in brain phosphocreatine (PCr) concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kondo, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes